CLINICAL TRIAL: NCT03532685
Title: Brazilian Severe Asthma Cohort Follow up: Clinical, Inflammatory and Functional Evaluation of a Population of Severe Asthmatics Based in Possible Phenotypes and Pathophysiologic Study of Obesity Association
Brief Title: Clinical, Inflammatory and Functional Evaluation of a Population of Severe and Obese Asthmatics: Follow up
Acronym: BRASAFUSP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Rafael Stelmach, Assistant Professor - Pulmonary Division - Heart Institute (InCor), University of Sao Paulo General Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: SDC - 4632/17/132; 82357517.0.0000.0068 (Other: Plataforma Brasil - Brazil Platform)
Record Dates: First submitted 2018-04-30; First posted 2018-05-22 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Severe Asthma; Obesity
Keywords: Asthma; severity; follow up; obesity; bariatric surgery
MeSH Terms: conditions — Asthma; Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Severe Asthma Obese Patients Surgery (Active Comparator): Bariatric surgery
  Interventions: Procedure: Bariatric
- Severe Asthma Obese Patients (No Intervention): usual care
- Severe Obese Patients (No Intervention): usual care

INTERVENTIONS:
Procedure: Bariatric — withdrawing a part of the stomach and may or may not be combined with bowel deviation
  Arms: Severe Asthma Obese Patients Surgery

SUMMARY:
In the study of a population of severe asthmatics, not controlled despite the treatment conducted, it was possible to evidence 5 phenotypic groups of patients. According to the refractoriness of the response to treatment, severe asthma may be phenotype in some distinct groups.Other prospective study found a large proportion of severe asthmatics with persistent airway obstruction, despite optimized treatment and systematic follow-up. Small airway involvement and remodelling, characterized by bronchial muscle thickening, appear to be the main culprits for asthma severity and persistent obstruction in this population.A point of interest in the severe asthmatics cohort was the vast majority were female and there were a considerable number of obese. Recent reviews show that the more consistent division of phenotypes in patients with severe asthma is still based on 3 previously described criteria (presence of atopy, eosinophilia and age of onset of asthma) and a more recent criterion for the presence of multi-comorbidities. Heterogeneity is the rule, the presumption of a natural evolution of gravity is not confirmed and the overlap of clusters is frequent. The stability and natural history of the phenotypes is poorly understood, postulating that the inflammatory activation of the severe asma is multifactorial and may resemble that described in the oncology literature.To date, there are no markers that allow prediction of lung evolution of most patients with severe asthma, and which patients are at greater risk of developing persistent or accelerated loss airflow or lung function, factors determining the severity of asthma. It is also unclear whether and how much phenotype-based treatment impact on disease control and prognosis. Future studies will be instrumental in defining how and why. These phenotypes are evolving, leading to the disabling characteristics of severe asthma and what may be the more effective therapeutic approaches for these patients. Since the initiated research group from 2006 has an extensive clinical, functional, inflammatory, tomographic and morphological evaluation of a cohort of patients with severe asthma, the ideal scenario exists to advance the understanding and investigation of the evolution of this rare disease through standardized follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe asthma (GINA step 3-5), followed in the outpatient clinic
* Non-smokers, smokers or former smokers of ≤ 10 packets per year. For smokers, <10 cigarettes / day and with onset asthma before onset of smoking
* Obese asthma patients BMI>30 kg / m2 FEV1 pre bronchodilator between 50 and 80% predicted
* Normal Chest Xray

Exclusion Criteria:

* Pregnancy
* Patients with a history of neoplasia, HIV + or other comorbidities that may interfere in the the study
* Patients with no understanding of the study procedures or who are not able to give their free and informed consent;
* Patients with other lung diseases such as chronic obstructive pulmonary disease, bronchiectasis, cystic fibrosis, or other lung diseases that may interfere with the study evaluation;
* Non adherence to standard asthma treatment;
* Inability to perform lung function assessment tests;
* Pulmonary exacerbation up to 30 days before the first study evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2018-05 (Estimated); Primary Completion 2018-05 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Forced Expiratory Volume first second (FEV1) - Unit: liters | up to 10 years
  To assess the rate of loss of lung function in patients with severe asthma, who remain in regular follow - up and under adequate therapy since 2006.
Impulse oscillometry: combined resistance and reactance measures (R5, R20, R5-20) kilopascal - unit: Liters -1/second -1 | 6-8 months
  To evaluate the functional airways characteristics of obese asthmatic patients, compared to non-obese asthmatics, before and after bariatric surgery

SECONDARY OUTCOMES:
Asthma exacerbations - unit: exacerbation/patient/year (number) | up to 10 years
  Rate of exacerbations per patient/year
Bronchial thickening measures overtime - unit: Percentage (%) bronchial wall area | up to 10 years
  To compare the degree of bronchial thickening, through chest tomography
Morbimortality - unit: number patients/year | up to 10 years
  Mortality and Hospitalizations per patient/year
Residual Volume (RV) - Liters | uo to 10 years
  To compare the degree of air trapping
Total Lung Capacity (TLC) - Liters | up to 10 years
  To compare the degree of air tapping
Ratio Residual Volume/Total Lung Capacity - Percentual (%) | up to 10 years
  To compare the degree of air trapping
Nitrogen Washout Test - Percentual (%) | up to 10 years
  To compare the heterogeneity amount of small airways

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Cukier, M/D, Study Director — Unversity of Sao Paulo - Pulmonary Division

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Carvalho-Pinto RM, Cukier A, Angelini L, Antonangelo L, Mauad T, Dolhnikoff M, Rabe KF, Stelmach R. Clinical characteristics and possible phenotypes of an adult severe asthma population. Respir Med. 2012 Jan;106(1):47-56. doi: 10.1016/j.rmed.2011.08.013. Epub 2011 Sep 3. PMID 21890336
- [Result] Carvalho-Pinto RM, Agondi RC, Giavina-Bianchi P, Cukier A, Stelmach R. Omalizumab in patients with severe uncontrolled asthma: well-defined eligibility criteria to promote asthma control. J Bras Pneumol. 2017 Nov-Dec;43(6):487-489. doi: 10.1590/S1806-37562017000000012. No abstract available. PMID 29340498
- [Result] Ferreira DS, Carvalho-Pinto RM, Gregorio MG, Annoni R, Teles AM, Buttignol M, Araujo-Paulino BB, Katayama EH, Oliveira BL, Del Frari HS, Cukier A, Dolhnikoff M, Stelmach R, Rabe KF, Mauad T. Airway pathology in severe asthma is related to airflow obstruction but not symptom control. Allergy. 2018 Mar;73(3):635-643. doi: 10.1111/all.13323. Epub 2017 Oct 23. PMID 28960335
- [Result] Ferreira PG, Freitas PD, Silva AG, Porras DC, Stelmach R, Cukier A, Fernandes FLA, Martins MA, Carvalho CRF. Dynamic hyperinflation and exercise limitations in obese asthmatic women. J Appl Physiol (1985). 2017 Sep 1;123(3):585-593. doi: 10.1152/japplphysiol.00655.2016. Epub 2017 Jul 6. PMID 28684597
- [Result] Athanazio R, Carvalho-Pinto R, Fernandes FL, Rached S, Rabe K, Cukier A, Stelmach R. Can severe asthmatic patients achieve asthma control? A systematic approach in patients with difficult to control asthma followed in a specialized clinic. BMC Pulm Med. 2016 Nov 16;16(1):153. doi: 10.1186/s12890-016-0314-1. PMID 27852260
- [Result] Freitas PD, Ferreira PG, da Silva A, Trecco S, Stelmach R, Cukier A, Carvalho-Pinto R, Salge JM, Fernandes FL, Mancini MC, Martins MA, Carvalho CR. The effects of exercise training in a weight loss lifestyle intervention on asthma control, quality of life and psychosocial symptoms in adult obese asthmatics: protocol of a randomized controlled trial. BMC Pulm Med. 2015 Oct 21;15:124. doi: 10.1186/s12890-015-0111-2. PMID 26487563
- [Result] Dias-Junior SA, Reis M, de Carvalho-Pinto RM, Stelmach R, Halpern A, Cukier A. Effects of weight loss on asthma control in obese patients with severe asthma. Eur Respir J. 2014 May;43(5):1368-77. doi: 10.1183/09031936.00053413. Epub 2013 Nov 14. PMID 24232701